CLINICAL TRIAL: NCT06742476
Title: Effectiveness Of Apneic Oxygenation During Induction Of General Anesthesia In Children Undergoing Adenotonsillectomy (As Partially Obstructed Airway)
Brief Title: Effectiveness Of Apneic Oxygenation During Induction Of General Anesthesia In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Safaa Gaber Ragab, Associate professor of anaesthiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: M738
Record Dates: First submitted 2024-12-12; First posted 2024-12-19 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction | interventions — Cannula

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Patients in the group A will undergo tracheal intubation without apneic oxygenation
- apniec oxygenation group (Experimental): Patients in the group B will undergo tracheal intubation in addition to apneic oxygenation at a flow 0.2 mg/kg using nasal cannula
  Interventions: Device: nasal cannula

INTERVENTIONS:
Device: nasal cannula — In the apneic oxygenation group, nasal cannula will be employed to administer continuous oxygenation, utilizing a flow rate of 0.2 L/kg, during the apneic phase while tracheal intubation is performed. Successful intubation will be confirmed by auscultation and the appearance of a square wave capnogragh.
  Arms: apniec oxygenation group

SUMMARY:
During general anesthesia, the administration of anesthetics and muscle relaxants induces apnea, wherein spontaneous breathing ceases . Pediatric patients, characterized by their higher oxygen consumption rate and smaller functional residual capacity, are particularly susceptible to hypoxemia during apneic episodes . This vulnerability to hypoxemia underscores the critical need for effective oxygenation strategies during anesthesia. Apneic oxygenation, the provision of oxygen without concurrent tidal volume delivery, emerges as a vital technique in pediatric anesthesia, playing a pivotal role in both routine and challenging airway management scenarios .

In modern practice, apneic oxygenation during airway management denotes the uninterrupted supply of oxygen, extending the window for maintaining safe oxygen saturation levels during the apneic phase . This technique holds particular significance in pediatric patients undergoing adenotonsillectomy, where the delicate balance of oxygenation is paramount .

Adenotonsillectomy, a common surgical procedure in pediatric patients, poses unique challenges in airway management . The procedure involves the removal of the adenoids and tonsils, often necessitating general anesthesia and temporary airway obstruction . Furthermore, the potential for blood and secretions in the oropharynx increases the risk of airway compromise during the perioperative period. In this context, ensuring adequate oxygenation is essential to mitigate the risk of hypoxemia and its associated complications In this randomized clinical trial, the investigators aim to evaluate the efficacy and safety of apneic oxygenation using nasal cannula in pediatric patients undergoing adenotonsillectomy under general anesthesia. By assessing our primary outcome and secondary outcomes, the investigators seek to contribute valuable insights into optimizing anesthesia management protocols for this vulnerable patient population.

DETAILED DESCRIPTION:
Following permission from the local institutional review board and institutional ethics committee, this study will be carried out at the FAYOUM University hospital. The research will employ a single -blinded, randomized, and controlled approach.

Prior to recruitment and randomization, detailed consent will be obtained from the parents or legal guardians of eligible patients.

Patients were randomly allocated 1: 1 to the two study groups:

Group (A):

Patients in the group A will undergo tracheal intubation without apneic oxygenation

Group (B):

Patients in the group B will undergo tracheal intubation in addition to apneic oxygenation at a flow 0.2 mg/kg using nasal cannula The randomization will be computer generated random number and the randomization sequence will be kept hidden in sealed opaque envelopes just opened after recruitment and admittance to the operating room. The group's allocations will be only blinded to parents of children.

In both the control and experimental groups, subjects will undergo a standardized general anesthesia protocol. All pediatric participants will receive premedication in the form of 0.5 mg/kg rectal midazolam upon admission to the operating theater, patients will be comfortably positioned on the operating table. Standard monitoring devices, including electrocardiography (ECG), non-invasive blood pressure (NIBP) measurement, pulse oximetry, and end-tidal carbon dioxide (EtCO2) monitoring, will be affixed. Intravenous access will be established to facilitate fluid and medication administration. In instances where venous access proves challenging, patients will be induced with inhaled sevoflurane at 8% concentration, followed by the insertion of an intravenous cannula. Subsequently, anesthetic induction will be achieved using a combination of 2 - 3 mg/kg of Propofol, 1 mcg/kg of Fentanyl, and 0.5 mg/kg of Atracurium. Following induction, bag-mask ventilation with 100% oxygen and flow rates of 6-8 litres min will be initiated for 3 minutes Ventilation will then be discontinued. In the apneic oxygenation group, nasal cannula will be employed to administer continuous oxygenation, utilizing a flow rate of 0.2 L/kg, during the apneic phase while tracheal intubation is performed. Successful intubation will be confirmed by auscultation and the appearance of a square wave capnogragh.

Following intubation, SpO2 levels will be recorded, and mechanical ventilation will be instituted to maintain normocapnia and oxygenation within predetermined target ranges.

In case of desaturation, the procedure will be discontinued as soon as the SpO2 reach 92%. Bag mask ventilation with 100% oxygen will be started until spo2 reach 100%, Intubation will then be performed by the supervising consultant anesthesiologist

ELIGIBILITY:
Inclusion Criteria:

* Patients (3 - 10 Years).
* Patients who were scheduled for adenotonsillectomy.
* ASA I and II

Exclusion Criteria:

* When nasal intubation is needed.
* Patients reported with nasal obstruction.
* Patients with any respiratory disease like asthma or recent upper respiratory tract infection.
* Patients with obstructive sleep apnea
* Patients with congenital heart disease
* Patients suspected difficult intubation or syndromatic patients eg : down syndrome , Goldenhar Syndrome , Pierre Robin syndrome … etc

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Lowest oxygen saturation during tracheal intubation. | at the end of intubation procedure
  Following intubation, SpO2 levels will be recorded

SECONDARY OUTCOMES:
Number of patients that their spo2 dropped to 95%. | at the end of intubation procedure
Number of patients that their spo2 dropped to 92%. | at the end of intubation procedure
Number of patients that their spo2 dropped to below 92%. | at the end of intubation procedure
Spo2 base line Spo2 after bag and mask ventillation and Spo2 immediately after intubation. | at the end of intubation procedure
Number of intubation attempts. | at the end of intubation procedure
Time of intubation. | at the end of intubation procedure
Number of patients developed bradycardia. | at the end of the study ( 6 months )

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Gaber Ragab, MD, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhananker SM, Ramamoorthy C, Geiduschek JM, Posner KL, Domino KB, Haberkern CM, Campos JS, Morray JP. Anesthesia-related cardiac arrest in children: update from the Pediatric Perioperative Cardiac Arrest Registry. Anesth Analg. 2007 Aug;105(2):344-50. doi: 10.1213/01.ane.0000268712.00756.dd. PMID 17646488
- [Background] van Munster JJCM, Zamanipoor Najafabadi AH, Schoones JW, Peul WC, van den Hout WB, van Benthem PPG. The impact of new evidence on regional variation in paediatric tonsillectomy and adenoidectomy: a historical review. J Laryngol Otol. 2020 Dec;134(12):1036-1043. doi: 10.1017/S002221512000273X. PMID 33431080
- [Background] Noda M, Shimada MD, Koshu R, Saito C, Ito M. Efficacy of endoscopic powered intracapsular tonsillectomy and adenoidectomy for pediatric obstructive sleep apnea: A retrospective case-control study. Auris Nasus Larynx. 2023 Jun;50(3):383-388. doi: 10.1016/j.anl.2022.08.008. Epub 2022 Sep 7. PMID 36085267
- [Background] Randall DA. Current Indications for Tonsillectomy and Adenoidectomy. J Am Board Fam Med. 2020 Nov-Dec;33(6):1025-1030. doi: 10.3122/jabfm.2020.06.200038. PMID 33219085
- [Background] Soneru CN, Hurt HF, Petersen TR, Davis DD, Braude DA, Falcon RJ. Apneic nasal oxygenation and safe apnea time during pediatric intubations by learners. Paediatr Anaesth. 2019 Jun;29(6):628-634. doi: 10.1111/pan.13645. Epub 2019 Apr 29. PMID 30943324
- [Background] Olayan L, Alatassi A, Patel J, Milton S. Apnoeic oxygenation by nasal cannula during airway management in children undergoing general anaesthesia: a pilot randomised controlled trial. Perioper Med (Lond). 2018 Feb 21;7:3. doi: 10.1186/s13741-018-0083-x. eCollection 2018. PMID 29484172
- [Background] Lyons C, Callaghan M. Uses and mechanisms of apnoeic oxygenation: a narrative review. Anaesthesia. 2019 Apr;74(4):497-507. doi: 10.1111/anae.14565. Epub 2019 Feb 19. PMID 30784037
- [Background] Kleine-Brueggeney M, Grosshauser M, Greif R. Apneic oxygenation in pediatric anesthesia. Curr Opin Anaesthesiol. 2022 Jun 1;35(3):361-366. doi: 10.1097/ACO.0000000000001127. PMID 35671025
- [Background] Nimmagadda U, Salem MR, Crystal GJ. Preoxygenation: Physiologic Basis, Benefits, and Potential Risks. Anesth Analg. 2017 Feb;124(2):507-517. doi: 10.1213/ANE.0000000000001589. PMID 28099321
- [Result] Tiradentes TAA, Einav S, Braz JRC, Nunes-Nogueira VS, Betini M, Corrente JE, Braz MG, Braz LG. Global anaesthesia-related cardiac arrest rates in children: a systematic review and meta-analysis. Br J Anaesth. 2023 Nov;131(5):901-913. doi: 10.1016/j.bja.2023.08.023. Epub 2023 Sep 22. PMID 37743151